CLINICAL TRIAL: NCT06244485
Title: A Phase 1b, Multicenter, Open-Label Study of Valemetostat Tosylate in Combination With DXd ADCs in Subjects With Solid Tumors
Brief Title: A Study of Valemetostat Tosylate in Combination With DXd ADCs in Subjects With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS3201-324
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumor; Valemetostat tosylate; DXD Antibody-drug Conjugates
MeSH Terms: interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: Dose Escalation Phase (Sub-protocol B) (Experimental): Participants with previously treated, advanced, or metastatic HER2-positive gastric or gastro-esophageal junction (GEJ) adenocarcinoma will receive valemetostat in combination with T-DXd.
  Interventions: Drug: Valemetostat tosylate; Drug: T-DXd
- Part 1: Dose Escalation Phase (Sub-protocol C) (Experimental): Participants with previously treated, locally advanced, unresectable, or metastatic non-squamous non-small cell lung cancer (NSCLC) with or without actionable genomic alteration(s) will receive valemetostat in combination with datopotamab deruxtecan (Dato-DXd).
  Interventions: Drug: Valemetostat tosylate; Drug: Dato-DXd
- Part 1: Dose Escalation (Sub-protocol A) (Experimental): Participants with unresectable or metastatic HER2-low IHC]1+ or IHC 2+/ISH-negative breast cancer will receive valemetostat in combination with T-DXd.
  Interventions: Drug: Valemetostat tosylate; Drug: T-DXd
- Part 2: Dose Expansion (Sub-protocol B) (Experimental): Participants with previously treated, advanced, or metastatic HER2-positive gastric or gastro-esophageal junction (GEJ) adenocarcinoma will receive valemetostat at the RDE in combination with T-DXd at RDE.
  Interventions: Drug: Valemetostat tosylate; Drug: T-DXd
- Part 2: Dose Expansion (Sub-protocol C) (Experimental): Participants with previously treated, locally advanced, unresectable, or metastatic non-squamous non-small cell lung cancer (NSCLC) with or without actionable genomic alteration(s) will receive valemetostat at the RDE in combination with datopotamab deruxtecan (Dato-DXd).
  Interventions: Drug: Valemetostat tosylate; Drug: Dato-DXd
- Part 2: Dose Expansion (Sub-protocol A) (Experimental): Participants with unresectable or metastatic HER2-low IHC]1+ or IHC 2+/ISH-negative breast cancer will receive valemetostat at the RDE in combination with T-DXd at RDE.
  Interventions: Drug: Valemetostat tosylate; Drug: T-DXd

INTERVENTIONS:
Drug: Valemetostat tosylate — Administered orally once daily
  Other Names: DS-3201b
Drug: T-DXd — One IV infusion Q3W on Day 1 of each 21-day cycle
  Other Names: DS-8201a; ENHERTU
  Arms: Part 1: Dose Escalation (Sub-protocol A); Part 1: Dose Escalation Phase (Sub-protocol B); Part 2: Dose Expansion (Sub-protocol A); Part 2: Dose Expansion (Sub-protocol B)
Drug: Dato-DXd — One IV infusion Q3W on Day 1 of each 21-day cycle.
  Other Names: DS-1062a
  Arms: Part 1: Dose Escalation Phase (Sub-protocol C); Part 2: Dose Expansion (Sub-protocol C)

SUMMARY:
This study will evaluate the safety, tolerability, and efficacy of valemetostat tosylate in combination with DXd ADC in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a 2-part study of valemetostat in combination with DXd ADCs in patients with HER2-positive gastric cancer, non-squamous NSCLC, or unresectable or metastatic HER2 low breast cancer. The study will begin with a Part 1 Dose-escalation Phase and will continue until the recommended dose for expansion "RDE" of valemetostat is determined and will then be followed by a Part 2 Dose-expansion Phase to further evaluate the safety and tolerability of the combination.

ELIGIBILITY:
Key Inclusion Criteria

All participants must meet all of the following criteria, as well as all criteria from the relevant sub-protocol to be eligible for enrollment:

* At least 18 years or the minimum legal adult age (whichever is greater) at the time the ICF is signed.
* Has at least 1 measurable lesion based on investigator imaging assessment (computed tomography or magnetic resonance imaging) using RECIST v 1.1 at Screening.
* Is willing to provide an adequate tumor sample.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1 at Screening.

Additional Key Inclusion for Sub-Protocol A:

* Diagnosed with pathologically documented breast cancer that:

  1. Is unresectable or metastatic.
  2. Has progressed on and would no longer benefit from endocrine therapy in hormone receptor-positive subjects in the opinion of the investigator.
  3. Has been treated with at least 1 and at most 2 prior lines of chemotherapy in the recurrent or metastatic setting.
  4. Has a history of low HER2 expression, defined as IHC 2+ /ISH-negative or IHC 1+ (ISH-negative or untested). ), as classified by the American Society of Clinical Oncology/College of American Pathologists 2018 HER2 testing guidelines.
  5. Was never previously HER2-positive (IHC 3+ or IHC 2+/ISH+) on prior pathology testing (per American Society of Clinical Oncology/College of American Pathologists guidelines

     Additional Key Inclusion for Sub-Protocol B:

     • Gastric or GEJ adenocarcinoma that is (a) unresectable or metastatic or (b) has progressed on trastuzumab or approved trastuzumab biosimilar-containing regimen.

     Additional Key Inclusion for Sub-Protocol C:
* Pathologically documented Stage IIIB, IIIC, or IV non-squamous NSCLC with or without AGA at the time of enrollment.
* Must meet prior therapy requirements:

  * Participants without AGA: (a) received platinum-based chemotherapy in combination with α-PD-1/α -PD-L1 mAb as a prior line of therapy or (b) received platinum-based chemotherapy and α -PD-1/ α -PD-L1 mAb (in either order) sequentially as 2 prior lines of therapy.
  * Participants with AGA: (a) has been treated with at least 1 or 2 prior lines of applicable targeted therapy that is locally approved for participant's genomic alteration at the time of Screening, (b) participants who have received platinum-based chemotherapy as a prior line of cytotoxic therapy, (c) may have received α -PD-1/α -PD-L1 mAb alone or in combination with a cytotoxic agent

Key Exclusion Criteria

* Has previously been treated with any enhancer of zeste homolog inhibitors.
* Uncontrolled or significant cardiovascular disease.
* Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.
* Has leptomeningeal carcinomatosis or metastasis.
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses.
* Current use of moderate or strong cytochrome P450 (CYP)3A inducers.
* Systemic treatment with corticosteroids (>10 mg daily prednisone equivalents).
* History of severe hypersensitivity reactions to other monoclonal antibodies (mAbs).
* Evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection requiring treatment with intravenous (IV) antibiotics, antivirals, or antifungals.
* Female who is pregnant or breastfeeding or intends to become pregnant during the study.
* Psychological, social, familial, or geographical factors that would prevent regular follow-up.

Additional Key Exclusion for Sub-Protocol A:

* Has previously received any anti-HER2 therapy in the metastatic setting.
* Has received prior treatment with an antibody-drug conjugate that consists of an exatecan derivative that is a topoisomerase I inhibitor, including either as part of prior treatment history or within prior participation in a clinical study.

Additional Key Exclusion for Sub-Protocol B:

* Participants who have received an antibody-drug conjugate consisting of an exatecan derivative that is a topoisomerase I inhibitor.

Additional Key Exclusion for Sub-Protocol C:

* Has received any agent, including an ADC, containing a chemotherapeutic agent targeting topoisomerase I or TROP2-targeted therapy including Dato-DXD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting Dose-limiting Toxicities (Part 1 Dose Escalation) | Cycle 1 Day 1 up to Day 21 (each cycle is 21 days)
Number of Participants Reporting Treatment-emergent Adverse Events (Part 1 Dose Escalation) | Screening up to 40 days after last dose
Objective Response Rate Based on Investigator Assessment (Part 2 Dose Expansion) | Baseline (Screening), at every 6 weeks from Cycle 1 Day 1 in the first year, and every 12 weeks thereafter until disease progression or until the start of a new anticancer treatment, up to approximately 5 years
  Objective response rate (ORR) is defined as the proportion of participants with a best overall response of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST v 1.1 criteria. CR is defined as a disappearance of all target lesions and PR is defined as at least a 30% decrease in the sum of diameters of target lesions.

SECONDARY OUTCOMES:
Overall Survival | Date of enrollment up to date of death due to any cause, up to approximately 5 years
Progression-free Survival | Date of enrollment up to date of radiographic disease progression or death due to any cause (whichever occurs first), up to approximately 5 years
  Disease progression will be determined by investigator assessment of tumor scans and using RECIST v 1.1 criteria.
Duration of Response (DoR) | Date of first documentation of objective tumor response (CR or PR) that is subsequently confirmed to the first documentation of objective tumor progression or to death due to any cause (whichever occurs first), up to approximately 5 years
  CR is defined as a disappearance of all target lesions and PR is defined as at least a 30% decrease in the sum of diameters of target lesions.
Objective Response Rate Based on Investigator Assessment (Part 1 Dose Escalation) | Baseline (Screening), at every 6 weeks from Cycle 1 Day 1 in the first year, and every 12 weeks thereafter until disease progression or until the start of a new anticancer treatment, up to approximately 5 years
  Objective response rate (ORR) is defined as the proportion of participants with a best overall response of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST v 1.1 criteria. CR is defined as a disappearance of all target lesions and PR is defined as at least a 30% decrease in the sum of diameters of target lesions.
Number of Participants Reporting Treatment-emergent Adverse Events (Part 2 Dose Expansion) | Screening up to 40 days after last dose
Total and Unbound Plasma Concentration of Valemetostat | Cycle 1, Day 1: Predose, 1 hour (hr), 2 hr, 4 hr, and 5 hr postdose; Cycle 1, Day 8 and Day 15: Predose; Cycles 2, 3, 4, Day 1: Predose (each cycle is 21 days)
Plasma Concentration of DXd Antibody-Drug Conjugates | Cycle 1, Day 1: Predose, 1 hour (hr), 2 hr, 4 hr, and 5 hr postdose; Cycle 1, Day 8 and Day 15: Predose; Cycles 2, 3, 4, Day 1: Predose (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (38):
- United States (20):
  - City of Hope At Orange County Lennar Foundation Cancer Center, Irvine, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - Brcr Medical Center, Inc Dba Boca Raton Clinical Research, Plantation, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Inc, Tampa, Florida
  - University of Hawaii At Manoa, Honolulu, Hawaii
  - University of Chicago Medical Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center (Mskcc) - New York, New York, New York
  - Clinical Research Alliance, Westbury, New York
  - Unc Hospitals, Chapel Hill, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - Ut Southwestern Medical Center, Dallas, Texas
  - University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Next Virginia, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- China (7):
  - Peking University Third Hospital, Beijing
  - Sun Yat-Sen University, Cancer Center, Guangzhou
  - SunYat-Sen University Cancer Center, Guangzhou
  - Harbin Medical Univeristy Cancer Hospital, Heilongjiang
  - Hunan Cancer Hospital, Hunan
  - Jilin Cancer Hospital, Jilin
  - Jinana Center Hosptial, Shandong
- IRCCS Istituto Scientifico Romagnolo Per, Cesena, Italy
- Japan (10):
  - National Cancer Center Hospital, Chūōku
  - National Hospital Org-Kyushu Cancer Center, Fukuoka
  - National Cancer Center Hospital East, Kashiwa
  - The Cancer Institute Hospital of Jfcr, Kōtoku
  - Aichi Cancer Center Hospital, Nagoya
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Ōsaka-sayama
  - Shizuoka Cancer Center, Shizuoka
  - Osaka University Hospital, Suita
  - Kanagawa Cancer Center, Yokohama

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/